CLINICAL TRIAL: NCT06647238
Title: Second Time's the Charm: Evaluation of Pharmacist Interventions in Lipid Management for Secondary Prevention
Brief Title: Evaluation of Pharmacist Interventions in Lipid Management for Secondary Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00118029
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-10

CONDITIONS: Hyperlipidemia; Coronary Artery Disease
Keywords: Pharmacist intervention; Hyperlipidemia treatment; secondary prevention of cardiovascular disease
MeSH Terms: conditions — Hyperlipidemias; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Control group will not directly interact with investigators. Will perform retrospective chart review only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacist Intervention (Experimental): Pharmacist review of patient chart and follow up visits to prescribe appropriate therapy for hyperlipidemia.
  Interventions: Other: Pharmacist Intervention in lipid therapy
- Control (No Intervention): Chart review only

INTERVENTIONS:
Other: Pharmacist Intervention in lipid therapy — Pharmacist intervention may include but is not limited to prescribing (statins, ezetimibe, bempedoic acid, PCSK9 inhibitors, etc.), patient education, and medication access.
  Arms: Pharmacist Intervention

SUMMARY:
The primary objective of this research project is to compare the effect of pharmacist interventions versus usual care in the implementation of guideline directed lipid lowering therapies for secondary prevention.

DETAILED DESCRIPTION:
Studies have shown prevention of cardiovascular adverse events is directly proportional to percent reduction in low-density lipoprotein (LDL). This evidence explains why LDL targets for secondary prevention have continued to be lowered. Cholesterol guidelines have been updated recently and encourage the use of multiple lipid lowering therapies, in addition to statins, for secondary prevention. However, these novel agents can be expensive and difficult to acquire, making prescribing challenging for providers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of coronary artery disease
* low-density lipoprotein (LDL) > 55
* Primary Care Physician at 1 of 6 identified clinics

Exclusion Criteria:

* Patients who are no longer an active patient of one of the internal medicine practices
* Patients whose cholesterol is managed by another practice
* Women of childbearing age/potential
* Patients residing in hospice/Long Term Care facilities
* End-stage liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kayla Marvin, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Cabarrus, Concord, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacist Intervention | Control
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist Intervention | Control | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.13 (12.53) | 74.3 (8.43) | 70.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 23 | 21 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 27 | 33 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 39 | 40 | 79
  Unknown or Not Reported | 0 | 0 | 0
CVD History [Count of Participants; unit: Participants]
  STEMI | 3 | 3 | 6
  NSTEMI | 5 | 13 | 18
  Ischemic stroke | 26 | 16 | 42
  Symptomatic PAD | 0 | 2 | 2
  Other | 14 | 20 | 34
Pertinent Past Medical History [Count of Participants; unit: Participants]
  Prior CABG/PCI | 10 | 27 | 37
  Diabetes | 30 | 25 | 55
  Hypertension | 36 | 38 | 74
  Chronic Kidney Disease | 17 | 19 | 36
  Chronic Heart Failure | 8 | 16 | 24
  Current Smoker | 8 | 3 | 11
LDL [Mean (Standard Deviation); unit: md/dL] | 88.36 (30.02) | 88.45 (34.03) | 88.41 (31.91)
History of Statin Intolerance [Count of Participants; unit: Participants] | 9 | 8 | 17
Baseline Treatment [Count of Participants; unit: Participants]
  High-intensity statin | 28 | 28 | 56
  Low or moderate-intensity statin | 8 | 6 | 14
  Ezetimibe | 8 | 7 | 15
  Bile Acid Sequestrant | 1 | 0 | 1
  Fish Oil | 2 | 0 | 2
  Fibrate | 1 | 0 | 1
  None | 3 | 2 | 5
  Other | 1 | 1 | 2
Insurance Type [Count of Participants; unit: Participants]
  Medicaid | 5 | 1 | 6
  Medicare | 25 | 34 | 59
  Commercial | 7 | 4 | 11
  Tricare | 0 | 0 | 0
  Self-pay | 0 | 0 | 0
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Meet Low-density Lipoprotein (LDL) at Goal (<55)
Description: patients with LDL within goal (<55) (yes/no)
Time Frame: Month 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist Intervention | Control
Number analyzed (Participants) | 40 | 40
Participants | 17 | 3
Statistical Analysis 1: Comparison: Pharmacist Intervention vs Control; Test type: Superiority; p < 0.001, Chi-squared

2. Secondary Outcome: Percent Change in Low-density Lipoprotein (LDL)
Description: Percent LDL reduction (will use baseline LDL and lowest LDL)
Time Frame: Baseline to end of study period up to Month 5
Measure: Mean (Standard Deviation); unit: percent of change in low-density lipopro
Arm/Group | Pharmacist Intervention | Control
Number analyzed (Participants) | 40 | 40
percent of change in low-density lipopro | -32.9 (0.24) | -6.8 (0.15)

3. Secondary Outcome: Number of Participants With Medications Initiated or Titrated
Description: Number of Medications initiated or titrated
Time Frame: Baseline to end of study period up to Month 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist Intervention | Control
Number analyzed (Participants) | 40 | 40
Participants
  Statin Adjustment | 10 | 3
  Ezetimibe Initiation | 18 | 1
  PCKS9i initiation | 6 | 0
  Fenofibrate initiation | 0 | 1

4. Secondary Outcome: Prevalence of Elevated Lipoprotein(a)
Description: Number of Subjects with Prevalence of elevated Lipoprotein(a)
Time Frame: Baseline to end of study period up to Month 5
Population: No patients in the control arm had lipoprotein(a) tested during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist Intervention | Control
Number analyzed (Participants) | 24 | 0
Participants | 7 | 0

ADVERSE EVENTS:
Time Frame: Month 5
Description: Not collected for this behavioral Intervention Clinical Trial
Arm/Group | Pharmacist Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT06647238/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT06647238/ICF_001.pdf